CLINICAL TRIAL: NCT02280603
Title: A Single-center, Active-controlled, Randomized, Double-blind, Proof of Concept Clinical Trial to Explore the Efficacy and Safety of DA-4001 After Topical Application in Male Patients With Androgenetic Alopecia
Brief Title: Clinical Trial to Explore the Efficacy and Safety of DA-4001 After Topical Application
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA4001_AGAP_POC
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DA-4001C (Experimental): DA-4001C is administered
  Interventions: Drug: DA-4001C
- 5% minoxidil (Active Comparator): 5% minoxidil is administered
  Interventions: Drug: 5% minoxidil

INTERVENTIONS:
Drug: DA-4001C — 1ml by topical application twice a day
  Arms: DA-4001C
Drug: 5% minoxidil — 1ml by topical application twice a day
  Other Names: minoxyl
  Arms: 5% minoxidil

SUMMARY:
This study is designed to explore the efficacy and safety of DA-4001 after topical application in male patients with androgenetic alopecia

Design : Randomized, double-blind, active-controlled study

Investigational Product : Finasteride, minoxidil

ELIGIBILITY:
Inclusion Criteria:

* Basic and specific(BASP) classification : basic type is M2 or C2 and specific type is V1,V2 or F1,F2

Exclusion Criteria:

* Evidence of hair loss other than androgenetic alopecia
* Use of finasteride, dutasteride within previous 12 months
* Use of minoxidil within previous 6 months
* Use of androgenic or anti-androgenic agents within previous 6 months
* Use of steroid agents for local application to scalp or systemic application within previous 1 month
* History of hair transplantation, scalp reduction
* Coronary artery disease, arrhythmia, congestive heart failure, valvular haert disease, angina pectoris

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in target area hair count per cm2 at week 24, as assessed by phototrichogram | baseline and week 24

SECONDARY OUTCOMES:
Change from baseline in target area hair count per cm2 at week 16, as assessed by phototrichogram | Baseline and week 16
Improvement rate of target area hair count per cm2 at week 16 and week 24, as assessed by phototrichogram | Baseline, week 16,and week24
Improvement rate of target area mean hair diameter at week 16 and week 24, as assessed by phototrichogram | Baseline, week 16, and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Hoon Kang, M.D, Ph.D, Principal Investigator — The catholic univ. of korea, St.Paul's hospital
Locations (1):
- Catholic Medical Center, Seoul, Dongdaemun-gu, South Korea